# Non-Interventional Study

#### B1851217

# Assessment of 13-valent pneumococcal conjugate vaccine effectiveness among people with HIV in the United States

# Statistical Analysis Plan

(SAP)

Version: 1.3

Author: PPD (PPD , Pfizer Inc, New York, NY, USA)

.

Date: 07-Dec-2023

# **TABLE OF CONTENTS**

| 1. AMENDMENTS FROM PREVIOUS VERSION(S) | 4 |
|---|---|
| 2. LIST OF ABBREVIATIONS | 7 |
| 3. RATIONALE AND BACKGROUND | 9 |
| 4. STUDY OBJECTIVES AND HYPOTHESES | 9 |
| 4.1. Primary Objectives | 9 |
| 4.2. Secondary Objectives | 9 |
| 5. RESEARCH METHODS | 9 |
| 5.1. Study Design | 9 |
| 5.2. Study Population | 10 |
| 5.2.1. Inclusion Criteria | 10 |
| 5.2.2. Exclusion Criteria | 11 |
| 5.2.3. Subgroups and Stratification | 11 |
| 5.3. Variables | 12 |
| 5.3.1. Effectiveness Endpoints | 12 |
| 5.3.2. Covariates | 13 |
| 5.3.3. Negative Controls | 18 |
| 5.4. Data Sources | 18 |
| 5.5. Treatment Labels | 18 |
| 5.6. Sample Size and Power Calculations | 19 |
| 5.7. Missing Data | 19 |
| 5.8. Statistical Methodology and Analyses | 19 |
| 5.8.1. General Considerations | 19 |
| 5.8.2. Index Date and Follow-up | 19 |
| 5.8.3. Minimum Sample Size Requirements | 20 |
| 5.8.4. Inverse Probability of Treatment Weighting for Time-Varying Exposures | 20 |
| 5.8.5. Assessment of Covariate Balance | 21 |
| 5.8.6. Incidence Rates | 21 |
| 5.8.7. Vaccine Effectiveness | 22 |
| 5.8.8. Assessment of Residual Confounding | 22 |
| 5.8.9. Eligibility, Demographic, Clinical and Exposure Characteristics | 23 |

| 5.8.10. Summaries of Study Outcomes | 24 |
|------------------------------------------------------------------|----|
| 5.8.11. Analysis of Study Objectives | 24 |
| 5.8.12. Analysis of Negative Control Outcomes and Exposure | 24 |
| 6. REFERENCES | 25 |
| 7. APPENDICES | 26 |
| 7.1. Appendix A: Table shells | 26 |
| 7.2. Appendix B: R Example Code | 26 |
| 7.2.1. Example Data Formats for First Event and Recurrent Events | 26 |
| 7.2.2. Code for Generating IPTW and IPCW | 27 |
| 7.2.3. Code for Incidence Rates | 27 |
| 7.2.4. Code for Standardized Differences | 28 |
| 7.2.5. Code for Cox Models | 29 |
| 7.3. Appendix C: Diagnosis and Procedure Codes Used in the Study | 30 |

# 1. AMENDMENTS FROM PREVIOUS VERSION(S)

| Version | Date | Changes | Rationale |
|---|---|---|---|
| 1.3 | 07-Dec-2023 | Added 'in the United<br>States' to the title | Reflect protocol amendment |
| 1.3 | 07-Dec-2023 | Added age group and<br>PPSV23 number of doses<br>as potential stratification<br>variables | Reflect protocol amendment |
| 1.3 | 07-Dec-2023 | Updated potential negative control outcomes | Reflect protocol amendment |
| 1.3 | 07-Dec-2023 | Updated opportunistic infections list | Reflect protocol amendment |
| 1.3 | 07-Dec-2023 | Study follow-up now<br>begins six months after<br>the first HIV-related<br>ICD-9-CM or ICD-10-<br>CM code | Reflect protocol amendment |
| 1.3 | 07-Dec-2023 | Removed requirement for six months of continuous enrollment before members' first HIV-related ICD-9-CM or ICD-10-CM code, updated inclusion start date and removed exclusion for individuals with evidence of ART therapy during baseline period | Reflect protocol amendment |
| 1.2 | 10-Aug-2023 | Updated to SOP template version 3.0 | |
| 1.2 | 10-Aug-2023 | Added alternate definition of outpatient | Reflect protocol amendment |

| | | candidiasis infection and NDC table | |
|---|---|---|---|
| 1.2 | 10-Aug-2023 | Added time-varying covariates for annual HIV viral load testing and annual CD4 cell count testing and their CPT codes. Added time-varying covariates for respiratory virus season. | Reflect protocol amendment |
| 1.2 | 10-Aug-2023 | Study follow-up now<br>begins 90 days after<br>index and at least 90 days<br>of continuous enrolment<br>in medical plans is added<br>to the inclusion criteria | Reflect protocol amendment |
| 1.2 | 10-Aug-2023 | The two outpatient HIV-<br>related codes are now no<br>more than 730 days apart | Reflect protocol amendment |
| 1.2 | 10-Aug-2023 | 90 instead of 30-day<br>intervals now used for the<br>analysis of RZV | Needed due to low numbers of patients vaccinated with RZV overall and in each interval |
| 1.2 | 10-Aug-2023 | Updated person-time<br>exclusion in Incidence<br>Rates subsection of 7.1<br>from 29 to 89 days | Needed to reflect the previous<br>update to the number of days<br>separating recurrent events<br>from 30 to 90 days |
| 1.2 | 10-Aug-2023 | Added a definition of overall SMD | Needed for reporting in output table |
| 1.2 | 10-Aug-2023 | Specified cluster robust<br>standard errors for the<br>95% confidence intervals<br>for the incidence rates<br>based on recurrent events<br>and updated R code | Needed to account for multiple events per patient |

| 1.2 | 10-Aug-2023 | Updated Payor categories in Table 5.2 | Previous categories did not accurately represent the values in the database |
|---|---|---|---|
| 1.2 | 10-Aug-2023 | Added text and reference<br>to potentially correct<br>main results for any bias<br>identified from the<br>negative control outcome | Needed to clarify the potential calculation that will be used |
| 1.1 | 2-Jun-2023 | The number of days used to separate pneumonia and candidiasis episodes to identify independent events was increased from 30 to 90 days. | Unrealistically high numbers of recurrent events were generated for several patients when using 30 days. It was therefore decided that 30 days may be insufficient time to recover from these infections in a HIV population. This decision was taken prior to generating incidence rates by vaccination status and prior to generating vaccine effectiveness results using recurrent events. |
| 1.1 | 2-Jun-2023 | Included the reporting of incidence rates annually and during the time periods of interest. | Added to explore potential changes over time. |
| 1.1 | 2-Jun-2023 | Specified that covariates imbalanced after weighting may be included in final weighted models. | Added to clarify the purpose of the assessment of covariate balance. |
| 1.1 | 2-Jun-2023 | Updated example code<br>for standardized<br>differences | Fixed error in code to match description. |
| 1.0 | 20-Mar-2023 | N/A. First version | N/A |

# 2. LIST OF ABBREVIATIONS

| Abbreviation | Definition |
|---|---|
| AG | Andersen-Gill |
| ART | Antiretroviral therapy |
| ATE | Average treatment effect |
| CI | Confidence interval |
| Cox-MSM | Marginal structural Cox models |
| CPT | Current procedural terminology® |
| CSF | Cerebrospinal fluid |
| HIV | Human immunodeficiency virus |
| HR | Hazard ratio |
| ICD-9-CM | International Classification of Diseases, Ninth<br>Revision, Clinical Modification |
| ICD-10-CM | International Classification of Diseases, Tenth<br>Revision, Clinical Modification |
| ICD-9-PCS | International Classification of Diseases, Ninth<br>Revision, Procedure Coding System |
| ICD-10-PCS | International Classification of Diseases, Tenth<br>Revision, Procedure Coding System |
| IPCW | Inverse probability of censoring weighting |
| IPD | Invasive pneumococcal disease |
| IPTW | Inverse probability of treatment weighting |
| NDC | National Drug Code |
| NI | Non-interventional |

| PCV | Pneumococcal conjugate vaccine |
|--------|-----------------------------------------------|
| PCV13 | 13-valent pneumococcal conjugate vaccine |
| PPSV23 | 23-valent pneumococcal polysaccharide vaccine |
| PLWH | People living with HIV |
| RZV | Recombinant zoster vaccine |
| SMD | Standardized mean differences |
| SVI | Social Vulnerability Index |
| VE | Vaccine effectiveness |

Note: in this document, any text taken directly from the non-interventional (NI) study protocol is *italicized*.

#### 3. RATIONALE AND BACKGROUND

People living with HIV (PLWH) are at increased risk of pneumococcal infections, but there is a lack of data on 13-valent pneumococcal conjugate vaccine (PCV13) vaccine effectiveness (VE) in PLWH.

The purpose of this study is to estimate PCV13 VE against pneumococcal disease in PLWH aged ≥18 years, overall and, if feasible, at 3, 5, and 7 years of follow-up. The primary outcomes of interest are invasive pneumococcal disease (IPD), pneumococcal pneumonia and all-cause pneumonia.

#### 4. STUDY OBJECTIVES AND HYPOTHESES

## 4.1. Primary Objectives

The primary objectives of this study are:

- Estimate vaccine effectiveness (VE) of PCV13 for invasive pneumococcal disease (IPD) among people living with HIV (PLWH) ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up
- Estimate VE of PCV13 for pneumococcal pneumonia among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up
- 3. Estimate VE of PCV13 for all-cause pneumonia among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up.

## 4.2. Secondary Objectives

The secondary objectives of this study are:

- Estimate VE of PCV13 for pneumococcal pneumonia or pneumonia with unspecified causes among PLWH ≥18 years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up
- Estimate VE of PCV13 for pneumonia with unspecified causes among PLWH≥18
  years of age, overall and, if feasible, at 3, 5, and 7 years of follow-up.

## 5. RESEARCH METHODS

## 5.1. Study Design

The VE study will be a retrospective cohort study using health care administrative claims and laboratory data.

PLWH will be identified using administrative claims and include individuals with at least one inpatient International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) or International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) code related to HIV (Appendix Table 7.1) or at least 2 outpatient ICD-9-CM or ICD-10-CM codes at least 30 days, but no more than 730 days, apart during January 1, 2014 and December 31, 2021. PLWH are required to have at least six months of continuous enrollment in one or more health plans and pharmacy benefits after their first HIV-related ICD-9-CM or ICD-10-CM code. These six months of continuous enrollment will be considered the baseline period, during which baseline covariates including demographics, comorbidities, and preventative care will be measured. The baseline period was also selected to minimize the number of outcome events that existing prior to or triggered an HIV diagnosis.

The date following the last date of the baseline period will be defined as the index date. The end of the study will occur on the last date that administrative claims data will be available, September 30, 2022.

# 5.2. Study Population

PLWH will be identified by ICD-9-CM or ICD-10-CM diagnosis codes (Appendix Table 7.1). Information provided by Komodo Health indicated that approximately 175,000 individuals meet the eligibility criteria.

All PLWH in the provided Komodo Health who meet the following criteria will be included in the analysis.

## 5.2.1. Inclusion Criteria

 HIV infection defined as at least one inpatient International Classification of Diseases, Ninth Revision, Clinical Modification (ICD-9-CM) or International Classification of Diseases, Tenth Revision, Clinical Modification (ICD-10-CM) code related to HIV (Appendix Table 7.1) or ≥2 outpatient ICD-9-CM or ICD-10-CM codes at least 30 days, but no more than 730 days, apart during January 1, 2014 and December 31, 2021

AND

 At least 18 years of age at the time of the first recording of HIV-related ICD-9-CM or ICD-10-CM code

AND

 At least six months of continuous enrollment in medical and pharmacy plans after the first HIV-related ICD-9-CM or ICD-10-CM code between January 1, 2014 and December 31, 2021. A gap of 30 days or less in enrollment will be allowed during this six month period.

## 5.2.2. Exclusion Criteria

Patients meeting the following criterion will not be included in the study:

 Evidence of PCV13 vaccination before the first HIV-related ICD-9-CM or ICD-10-CM code

All available data prior to first HIV-related ICD-9-CM or ICD-10-CM code will be used to assess evidence of PCV13 vaccination, however there is no minimum time requirement.

## 5.2.3. Subgroups and Stratification

Several stratified analyses will be conducted. PPSV23 is recommended for PLWH and feasibility data provided by Komodo suggest that one in four PWLH who received PCV13 during 2014-2015 also received PPSV23 within two years. Rather than censor or exclude individuals who receive PPSV23, we will calculate PCV13 VE among PWLH who have/have not received PPSV23 before and during the study period. The analysis may also be stratified by the number of PPSV23 doses, e.g. 0, 1, 2+.

Feasibility assessments from Komodo indicate that approximately 25% of PWLH have at least one CD4 cell count or percentage laboratory result available. Therefore, we will calculate PCV13 VE among the subset of PWLH who have a CD4 cell count during the baseline period or follow-up, and potentially stratify by CD4 category using the patient's lowest value during the study.

Additional VE stratifications by ART adherence during follow-up, year of HIV diagnosis, and age will be assessed for feasibility as well, as these affect patients' immune status and immune reconstitution. Due to possible waning of the VE and different lengths of follow-up by index year, VE stratification by year of HIV diagnosis will be restricted to the first 3 years of follow-up (0 to 1079 days).

The above subgroup analyses will be conducted if there are sufficient numbers of patients/ events to maintain patient de-identification (Section 5.8.3) and where the 95% confidence intervals (CI) for the VE estimates can be expected to exclude zero in the best case scenarios for the analyses, i.e. the highest expected VE estimate, the lowest expected censoring rate and at the maximum follow-up time. Table 5.1 provides precision estimates for IPD and all-cause pneumonia under different numbers of individuals available for the analysis. The following assumptions were used for the estimates:

- 32% of individuals received PCV13
- IPD incidence among PLWH is 183 cases per 100,000 population [1]
- All-cause pneumonia incidence among PLWH is 5,487 cases per 100,000 population
- VE for IPD due to any serotype is 22.5% [2, 3]
- VE for all-cause pneumonia is 15% [4]

- Annual censoring of individuals due to loss to follow-up or death is 4%
- Up to 97 months of follow-up

Survival and censoring times were simulated assuming exponential distributions. Vaccination status was modelled as a time-varying covariate [5]. Hazard ratios were assumed as 1-(VE/100). Simulations were run 100 to 200 times per scenario. Cox regression models were run on each simulated dataset to estimate the 95% CIs for the log HRs. Means were generated and exponentiated to obtain the 95% CIs for the VEs using (1- HR) x 100 and used to describe VE precision.

Table 5.1 Precision of PCV13 Vaccine Effectiveness Estimates for Invasive Pneumococcal Disease and All-Cause Pneumonia Subgroup Analyses

| | IPD<br>VE: 22.5% | | All-cause pneumonia<br>VE: 15% | |
|---|---|---|---|---|
| Number of individuals | Lower 95%<br>confidence<br>interval<br>estimate | Upper 95%<br>confidence<br>interval<br>estimate | Lower 95%<br>confidence<br>interval<br>estimate | Upper 95%<br>confidence<br>interval<br>estimate |
| 87,000 (N/2) | 6% | 37% | 11% | 18% |
| 58,000 (N/3) | 1% | 40% | 11% | 19% |
| 43,000 (N/4) | -5% | 41% | 10% | 20% |
| 35,000 (N/5) | -6% | 44% | 9% | 20% |
| 29,000 (N/6) | -9% | 46% | 9% | 20% |
| 22,000 (N/8) | -16% | 49% | 8% | 21% |

Table 5.1 shows that, under the current assumptions, 95% CIs for the IPD VE would still be expected to exclude 0% in subgroups with 58,000 individuals. For all-cause pneumonia the 95% CIs for the VE would still be expected to exclude 0 in subgroups with fewer than 22,000 individuals. Therefore, the study should have sufficient precision to address the study the objectives in several of the planned subgroups.

#### 5.3. Variables

#### 5.3.1. Effectiveness Endpoints

The outcomes of interest for the primary and secondary objectives are listed in Table 5.2.

Episodes separated by at least 90 days will be considered independent events. For claims that include pneumonia that are separated by <90 days, those claims will be collapsed into a single episode with a date of the initial diagnosis.

Table 5.2 Outcomes of Interest

| Outcome Type | Outcome | Definition |
|---|---|---|
| Primary | IPD | ICD-9-CM or ICD-10-CM codes listed in Appendix |
| outcomes | | Table 7.4 |
| | Pneumococcal | ICD-9-CM or ICD-10-CM codes listed in Appendix |
| | pneumonia | Table 7.4 |
| | All-cause pneumonia | ICD-9-CM or ICD-10-CM codes listed in Appendix |
| | | Table 7.4 |
| Secondary | Pneumococca1 | ICD-9-CM or ICD-10-CM codes listed in Appendix |
| outcomes | pneumonia or | Table 7.5 |
| | pneumonia with | |
| | unspecified causes | |
| | Pneumonia with | ICD-9-CM or ICD-10-CM codes listed in Appendix |
| | unspecified causes | Table 7.5 |
| Sensitivity | All-cause pneumonia | ICD-9-CM or ICD-10-CM codes listed in Appendix |
| analysis outcome | not associated with | Table 7.6 |
| | HIV | |

For combination diagnosis codes, (e.g., bacteremia + pneumococcus) for diagnoses in an inpatient setting patients must have all codes within the same admission. The latest date of the combination of diagnoses will be used as the diagnosis date. For diagnoses in an outpatient setting patients must have all codes within the same date.

#### 5.3.2. Covariates

The list of demographic and clinical characteristics considered for descriptive reporting, subgroups and inclusion as covariates in models for generating the propensity scores are provided in Table 5.3. The Komodo Health database will be source of all variables.

Patients will be considered to have a comorbidity or hospitalization during baseline if there was evidence of a diagnosis at any time during the baseline period. Evidence of comorbidities or hospitalization during follow-up will be considered as new diagnoses. Once diagnosed, patients will be considered diagnosed for the remainder of their follow-up. ART adherence during baseline and follow-up will be updated every 6 months (180 days) based on the data collected in that previous timeframe. For baseline annual physical exam and annual influenza vaccine, patients will be considered adherent (coded as 'Yes') if there was evidence of these events at any time during the baseline period. During the follow-up, patients will be considered adherent up to 365 days after the last event date.

For annual CD4 and viral load laboratory tests during baseline and follow-up, patients will be coded as 'Yes' up to 365 days after the last event date. For respiratory virus season during follow-up, patients will be coded as 'Yes' if the observation time is in October, November, December, January, February, March or April.

The baseline period for the assessment of covariates is the six months prior to the index date, i.e., no data prior to six months will be included.

Covariates used at baseline only will be considered time-fixed confounders. Covariates additionally or only used during follow-up will be considered time-varying confounders.

Categories may be collapsed, or covariates may be excluded from the propensity scores if models fail to converge.

Table 5.3 List of Covariates

| Variable | Operational Definition | Role | Time of Use |
|---|---|---|---|
| Age in years | Calculated as [year individual meets HIV | Descriptive | Baseline |
| | criteria] – [birth year] | (continuous and | |
| | Categorized as: 18-49, 50-64, 65-74, and ≥75 years | categorical) | |
| | | Covariate | |
| | As a subgroup, age will be categorized as 18-49, 50-64 and 65+ years | (categorical) | |
| | 18-49, 50-04 and 05+ years | Subgroup | |
| | | (categorical) | |
| Sex | Male, Female, Other/ Unknown | Descriptive, | Baseline |
| | | covariate | |
| Social | SVI characterizes resiliency of a community | Descriptive, | Baseline |
| Vulnerability | when faced by external pressures and | covariate | |
| Index (SVI) | stresses[6, 7]. SVI ranges from 0 to 100, | | |
| | where a value of 100 indicates the most vulnerable population. | | |
| | 3-digit zip codes will be translated to 3-digit<br>zip code tabulation areas, and SVI will be<br>calculated at the 3-digit zip code tabulation<br>area. | | |
| | Categorized as: low (lowest quartile), average (middle two quartiles) and high (highest quartile). | | |
| US region | Northeast, North Central, South, West,<br>Unknown | Descriptive, covariate | Baseline |

| Payor | Commercial, Dually eligible, Medicaid/CHIP, | Descriptive, | Baseline |
|---|---|---|---|
| | Medicare, Missing, Other | covariate | |
| Year of HIV | Calendar year of first HIV diagnosis code | Descriptive, | Baseline |
| diagnosis | 2014, 2015, 2016, 2017, 2018, 2019, 2020, | covariate, | |
| | 2021. | subgroup | |
| | When used as a subgroup year will be | | |
| | categorized as 2014, 2015-2016, 2017-2018, | | |
| | 2019-2021. | | |
| Alcoholism | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| | Appendix Protocol Annex Table 1.1 | covariate | follow-up |
| | Yes, No | | |
| Asplenia | CPT/Healthcare Common Procedure Coding | Descriptive, | Baseline and |
| | System (HCPCS), ICD-10-Procedure Coding | covariate | follow-up |
| | System (ICD-10-PCS), ICD-9-Procedure | | |
| | Coding System (ICD-9-PCS), ICD-9-CM, or | | |
| | ICD-10-CM codes listed in Protocol Annex | | |
| | Table 1.2 | | |
| Chronic heart | CPT/HCPCS, ICD-10-PCS, ICD-9-PCS, | Descriptive, | Baseline and |
| disease | ICD-9-CM, or ICD-10-CM codes listed in | covariate | follow-up |
| | Protocol Annex Table 1.4 | | |
| | Yes, No | | |
| Chronic kidney | CPT/HCPCS, ICD-10-PCS, ICD-9-PCS, | Descriptive, | Baseline and |
| disease and | ICD-9-CM, or ICD-10-CM codes listed in | covariate | follow-up |
| renal failure | Protocol Annex Table 1.5 | | |
| | Yes, No | | |
| Chronic liver | CPT/HCPCS, ICD-10-PCS, ICD-9-PCS, | Descriptive, | Baseline and |
| disease | ICD-9-CM, or ICD-10-CM codes listed in | covariate | follow-up |
| | Protocol Annex Table 1.6 | | |
| | Yes, No | | |
| Chronic lung | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| disease | Protocol Annex Table 1.7 | covariate | follow-up |
| | Yes, No | | |
| Asthma | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| | Protocol Annex Table 1.3 | covariate | follow-up |
| | Yes, No | | |
| Diabetes | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| mellitus | Protocol Annex Table 1.9 | covariate | follow-up |
| | Yes, No | | |
| Generalized | CPT/HCPCS, ICD-10-PCS, ICD-9-PCS, | Descriptive, | Baseline and |
| malignancy | ICD-9-CM or ICD-10-CM codes listed in | covariate | follow-up |
| | Annex Table 1.10 | | |
| Immunosuppres | PLWH will be considered on | Descriptive, | Baseline and |
| sive medications | immunosuppressive medications if: | covariate | follow-up |
| | 1) ≥1 NDC, HCPCS, or ICD-10-PCS code in | | |
| | Appendix Table 7.7 | | |

| | <ol> <li>≥ 1 NDC (using orals only) in Appendix</li> </ol> | | |
|---|---|---|---|
| | Table 7.7 where the daily dose is $\geq$ 20mg or | | |
| | prednisone or prednisone equivalent for a | | |
| | duration of ≥14 consecutive days | | |
| | Yes, No | | |
| Leukemia | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| | Protocol Annex Table 1.12 | covariate | follow-up |
| Multiple | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| myeloma | Annex Table 1.13 | covariate | follow-up |
| Nephrotic | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| syndrome | Protocol Annex Table 1.14 | covariate | follow-up |
| -, | Yes, No | | |
| Non-Hodgkin's | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| lymphoma | Protocol Annex Table 1.15 | covariate | follow-up |
| Organ transplant | CPT/HCPCS, ICD-10-PCS, ICD-9-PCS, | Descriptive, | Baseline and |
| Organ transplant | ICD-9-CM or ICD-10-CM codes listed in | covariate | follow-up |
| | Protocol Annex Table 1.16 | Covariate | Ionow-up |
| Sickle cell | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| disease or other | Protocol Annex Table 1.17 | covariate | follow-up |
| hemoglobinopat | Yes, No | Covariate | Ionow-up |
| hies | 165, 140 | | |
| Hepatitis B | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| ricpatitis D | Protocol Annex Table 2.1 | covariate | follow-up |
| | Yes, No | COVALIALE | Ionow-up |
| Hepatitis C | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| riepautis C | Protocol Annex Table 2.2 | covariate | follow-up |
| | Yes, No | Covariate | Ionow-up |
| Cigarette | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| smoking | Protocol Annex Table 1.7 | covariate | follow-up |
| SHOKING | Yes, No | COVALIALE | Ionow-up |
| Annual physical | CPT/HCPCS codes listed in Protocol Annex | Descriptive, | Baseline and |
| exam | Table 3.1 | covariate | follow-up |
| CAMII | Yes, No | COVALIALE | Ionow-up |
| Annual | CPT/HCPCS, ICD-10-PCS, ICD-9-PCS, or | Descriptive | Baseline and |
| influenza | | Descriptive, | follow-up |
| vaccine | NDC codes listed in Appendix Table 7.8 | covariate | 10110W-up |
| | Yes, No | <b>D</b> | D 1 |
| Any pneumonia | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline |
| infection | Appendix Table 7.4 | covariate | |
| | Yes, No | | |
| Any | Evidence of inpatient claim(s) | Descriptive, | Baseline and |
| hospitalization | Yes, No | covariate | follow-up |
| Hodgkin's | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| lymphoma | Protocol Annex 1.11 | covariate | follow-up |
| | Yes, No | 1 | |
| Opportunistic | ICD-9-CM or ICD-10-CM codes listed in | Descriptive, | Baseline and |
| infections | Protocol Annex Table 14 | covariate | follow-up |

| | Yes, No | | |
|---|---|---|---|
| | Note: In the analysis of all-cause pneumonia, pneumocystis jirovecii pneumonia codes are excluded from the follow-up. In the analysis of candidiasis negative control outcomes, candidiasis infection codes are excluded from the follow-up. | | |
| Antiretroviral | ART use will be identified by NDC codes | Descriptive, | Baseline and |
| treatment (ART) | listed in Appendix Table 7.2 | covariate,<br>subgroup | follow-up |
| adherence | Adherence will be measured as 'Proportion of days covered = (Number of days covered by any ART, excluding ritonavir and cobicistat) ÷ (total days)*100'[8] every six months | suogroup | |
| | Individuals with >80% of days covered will<br>be classified as 'adherent' and individuals<br>with ≤80% of days covered will be classified | | |
| | as 'non-adherent' [8]. Individuals without<br>ART information will be classified as<br>Missing. | | |
| | As a subgroup, ART adherence will calculated using the information over the entire follow-up. | | |
| CD4 cell count | Categorized as <200, 200-499, ≥500 cells/mm <sup>3</sup> | Descriptive,<br>subgroup | Baseline and<br>follow-up |
| PPSV23 | NDC and CPT codes listed in Appendix | Descriptive, | Before first |
| vaccination | Table 7.9 | subgroup | HIV<br>diagnosis, |
| | Yes, No. | | baseline and |
| | 0, 1, 2+ doses | | follow-up |
| Annual CD4 | CD4 laboratory tests will be identified by | Covariate | Baseline and |
| laboratory test | CPT codes listed in Appendix Table 7.11 | | follow-up |
| | Individuals who have at least one CD4 | | |
| | laboratory test performed during each year of | | |
| | follow-up | | |
| Annual viral | Yes, No | Covariate | Baseline and |
| load laboratory | Viral load laboratory tests will be identified<br>by CPT codes listed in Appendix Table 7.12 | Covariate | follow-up |
| test | by CF1 codes fisted in Appendix Table 7.12 | | Tonow-up |
| | Individuals who have at least one viral load<br>laboratory test performed during each year of | | |
| | follow-up | | |
| | Yes, No | | |

| Respiratory | Respiratory virus season occurs between | Covariate | Follow-up |
|---|---|---|---|
| virus season | October 1 and April 30 | | |
| | Yes, No | | |

### 5.3.3. Negative Controls

# Table 5.4 List of Negative Control Variables

| Variable | Operational Definition | Role | Time of Use |
|---|---|---|---|
| Recombinant zoster | NDC and CPT codes listed in Appendix | Negative | Follow-up |
| vaccine (RZV; | Table 7.10 | control | |
| Shingrix, | | exposure | |
| GlaxoSmithKline) | | | |
| May include, but not | ICD-9-CM and ICD-10-CM codes | Negative | Follow-up |
| limited to, candidiasis | listed in Protocol Annex Table 4.1 | control | |
| infection, all-cause | | outcomes | |
| diarrhea and | Candidiasis infection: evidence of an | | |
| accidental injury | antifungal treatment within 7 days of | | |
| | outpatient candidiasis ICD-9-CM or | | |
| | ICD-10-CM codes will be explored. | | |
| | NDC and CPT codes listed in Appendix | | |
| | Table 7.13 | | |

#### 5.4. Data Sources

The source of data for the VE study will be health care administrative claims and HIV-laboratory data provided by Komodo Health. Komodo Health uses artificial intelligence and data analytics to combine and link patient-level information from more than 150 payers in the United States, including Medicare, Medicaid, and Commercial plans. Currently, Komodo Health has patient-level data on approximately 325 million individuals and these data include inpatient and outpatient claims, pharmacy dispensing claims, provider specialty claims, and mortality information.

Komodo Health will provide administrative claims available during January 1, 2014 through September 30, 2022 for individuals who have at least one ICD-9-CM or ICD-10-CM code related to HIV (Appendix Table 7.1) or at least one antiretroviral (ART) medication dispensed (Appendix Table 7.2).

#### 5.5. Treatment Labels

Information on PCV13 vaccination status will continue to be collected on and after index date and will therefore be treated as a time-varying exposure. PLWH in the study will be assigned to 'PCV13 Vaccinated' or 'PCV13 Unvaccinated' according to their vaccination status by each person-time record during the follow-up. Individuals will be considered vaccinated from 14 days after their PCV13 vaccination date till the remainder of their follow-up.

National Drug Codes (NDC) and Current Procedural Terminology® (CPT) codes used to identify PCV13 receipt are listed in Appendix Table 7.3.

## 5.6. Sample Size and Power Calculations

The planned analyses do not involve hypothesis testing and sample size calculations are not applicable. However, we examined the precision of PCV13 vaccine effectiveness for IPD and all-cause pneumonia among people living with HIV at 36 months and 97 months (which was the maximum follow-up time available from feasibility assessments) after index. This was conducted for the 175,000 individuals expected in the overall analysis (Protocol Section 9.5) and for varying potential subgroup sizes (Section 5.2.3).

# 5.7. Missing Data

No imputation for missing values will be performed. Subject to patient counts (Section 5.8.3), missing or 'unknown' values will be reported and analyzed as separate categories and included in the totals.

## 5.8. Statistical Methodology and Analyses

#### 5.8.1. General Considerations

Descriptive statistics will be used to summarize variables. For categorical variables, the frequency and percentage of patients in each category will be presented. Percentages will be based on the total number of relevant patients, including those with 'unknown' or missing values. For continuous variables, data will be presented as means, standard deviations, medians, 25th and 75th percentiles, minimums and maximums. Continuous variables may be additionally categorized and analyzed as categorical variables.

No statistical hypotheses are specified and there will be no correction for multiple comparisons.

Time in years between two dates will be calculated as (end date – start date) + 1, divided by 365.25, unless otherwise specified.

All data analysis will be conducted in R, version 4.1.3 or later (R Foundation for Statistical Computing, Vienna, Austria).

# 5.8.2. Index Date and Follow-up

The date following the last date of the baseline period will be defined as the index date. The end of the study will occur on the last date that administrative claims data will be available, September 30, 2022.

For PLWH who receive PCV13 after their index date, we will include the time between their index date and the 13 days after their PCV13 vaccination date as unvaccinated follow-up time. Any outcomes occurring during this time will be counted as events in the unvaccinated

cohort. Follow-up that occurs 14 days after PCV13 vaccination will be defined as vaccinated follow-up time.

Unvaccinated (no PCV13) PLWH will be followed from their index date until the earliest occurrence of the following: 13 days after PCV13 vaccination, death, end of health plan enrollment, or end of study period. Vaccinated PLWH will be followed from 14 days after their PCV13 vaccination date or index date if they were vaccinated during the baseline period, until the earliest occurrence of the following: death, end of health plan enrollment, or end of study period.

## 5.8.3. Minimum Sample Size Requirements

In order to maintain patient de-identification, outcomes, covariates and subgroups will have at least 10 patients/ events in each category for inclusion in outputs.

# 5.8.4. Inverse Probability of Treatment Weighting for Time-Varying Exposures

Except for patients vaccinated more than 13 days before the end of the baseline period, exposure (vaccination) status will not be fixed at start of follow-up, with patients able to receive PCV13 during follow-up. Therefore, PCV13 will be considered a time-varying exposure. The values for some clinical characteristics may also change during the study period and values during baseline may be poor proxies for covariate values at the various points during the follow-up. Therefore, some covariates will be treated as time-varying confounders (Section 5.3.2).

Inverse probability of treatment weighting (IPTW) will be generated from predicted probabilities of vaccination status (propensity scores) to create pseudo-populations where any imbalances in the potential confounders by vaccination status are reduced. For the analyses of first events, stabilized weights will be generated for each patient for the baseline period and every 30 days from index during the follow-up until the earliest of the following: outcome, death, end of health plan enrollment or end of study period. For the analyses of recurrent events, stabilized weights will be generated for each patient for the baseline period and every 30 days from index during the follow-up until the earliest of the following: death, end of health plan enrollment or end of study period. This aims to make vaccination status independent of the measured confounders at each of the follow-up timepoints [9]. The weights will be used to estimate the average treatment effect (ATE). For the analysis of RZV, stabilized weights will be generated every 90 days instead of 30, due to the expected lower numbers of patients vaccinated with RZV overall and in each interval.

The numerators for the stabilized weights will be the estimated probability of a patient's observed vaccination status at timepoint given their prior vaccination status and time-fixed covariates. The denominators will be the estimated probability of a patient's observed vaccination status at the given timepoint given their prior vaccination status, time-fixed covariates and time-varying covariates. Numerators and denominators after vaccination will be set to 1 and the cumulative product of these ratios will be calculated, therefore IPT

weights after vaccination will be constant. Time-varying covariates will be lagged, i.e., within each 30-day (or 90-day for RZV) interval the vaccination status will be the status at the end of the interval, whereas the values for the covariates will be from the end of the previous interval. Cox proportional hazards models will be used to model the associations between vaccination status and the numerators and denominators.

It is possible that censoring may be informative, with patient characteristics associated with loss to follow-up. Therefore, patients who are censored may have different risks of the study outcomes than patients who are not censored. Inverse probability of censoring weighting (IPCW) will also be generated during the follow-up using the above methods for IPTW. These weights will be multiplied by the IPT weights to produce a new set of weights [9].

Distributions of the IPT, IPC and IPT\*IPC weights will be summarized by vaccination status. In the presence of extreme/outlier weights, stabilized weights may be truncated at the 1<sup>st</sup> and 99<sup>th</sup> percentiles for use in the Cox models for the outcomes. Although there is no formal definition of an extreme weight, the need for truncation will be judged based on the distributions and the potential effect on the interpretation of results [9].

Weights for first and recurrent events will be generated separately in datasets created for each study outcome; however, all weights will be derived without assessing their impact on the VE estimates. Weights will also be generated again in each of the subgroups. The weights will generated using the *ipwtm* function within the *ipw* R package [10]. Example R code is provided in Appendix 7.2.

## 5.8.5. Assessment of Covariate Balance

Standardized mean differences (SMD) will be calculated for the baseline period and every 30 days (or 90 days for RZV) since index for each of the covariates up to any PCV13 vaccination before and after the IPTW. Overall SMDs will be presented for each covariate before and after the IPTW (such as median and maximum values across the intervals with at least 100 patients vaccinated), as well as those at the end of each year of follow-up (at 360, 720, 1080, 1440, 1800, 2190, 2550, 2910 days). SMDs ≤0.1 will be considered as evidence of negligible imbalance. Variables with SMDs >0.1 after IPTW may be added to final weighted outcome models.

#### 5.8.6. Incidence Rates

Incidence rates will be reported using first episodes only and again after including recurrent episodes of the same type. Crude incidence rates and 95% CIs will be presented as episodes per 100,000 person-years by PCV13 vaccination status for each outcome overall as well as annually and during time periods of interest (0-3, 3-5 and 5-7 years).

For incidence rates based on first episodes only, the total unvaccinated person-time will be calculated as time from index date to the earliest of the following: outcome, 13 days after their PCV13 vaccination, death, end of health plan enrolment or end of study period. The

total vaccinated person-time will be calculated as time from 14 days after their PCV13 vaccination date or index date, if they were vaccinated more than 13 days before the end of the baseline period, to the earliest of the following: outcome, death, end of health plan enrolment or end of study period.

For incidence rates including recurrent episodes of the same type (separated by at least 90 days), the total unvaccinated person-time will be calculated as time from index date to the earliest of the following: 13 days after their PCV13 vaccination, death, end of health plan enrolment or end of study period. The total vaccinated person-time will be calculated as time from 14 days after their PCV13 vaccination date or index date, if they were vaccinated more than 13 days before the end of the baseline period ,to the earliest of the following: death, end of health plan enrolment or end of study period. Person-time will exclude any time the patient is not at risk, i.e. the first 89 days after an episode. Cluster robust standard errors will be used in the calculation of 95% confidence intervals to account for multiple events per patient.

#### 5.8.7. Vaccine Effectiveness

Crude PCV13 VE percentages will be estimated based on (1-HR) x 100, where HR is obtained from unadjusted Cox models for first episodes for each outcome. VE percentages will also be obtained from marginal structural Cox models (Cox-MSM) after applying the IPT and the IPT\*IPC weights. As the numerators for the stabilized weights will include the index-fixed covariates, those covariates will also be included in the Cox-MSM for the outcomes [9]. Cluster robust standard errors will be used to account for the multiple records per patient. The proportional hazards assumption will be assessed graphically with the inspection of Schoenfeld residuals.

To explore potential changes in VE over time, HRs may also be generated during specific time periods using piecewise Cox models. The time periods will be 0-3 years (0 to 1079 days), 3-5 years (1080 to 1799 days), 5-7 years (1800 to 2549 days).

VE may also be assessed for recurrent events using the Andersen-Gill (AG) model [11]. For each outcome, subsequent events will be of the same type, e.g., in the analysis of IPD it will be assumed that a patient is only at risk for future IPD events. The VE is assumed constant across the recurrent events.

#### 5.8.8. Assessment of Residual Confounding

Residual confounding of our VE estimates due to inadequate control for health care seeking behavior and immune status in our analyses will be explored. To do so, we will employ a negative control exposure and a negative control outcome. Potential negative control exposures include vaccinations that are recommended for PLWH but would not be expected to have any protective effect against the pneumonia outcomes of interest. We plan to use recombinant zoster vaccine (RZV) as the negative control exposure. Current US clinical guidelines recommend that PLWH be offered RZV vaccination. Therefore, we will develop a

model for our study population in which the exposure is at least one dose of RZV and the outcomes are our primary outcomes of interest. If residual confounding does not exist, RZV would not have an effect on the pneumonia outcomes. However, if the analysis demonstrates that RZV protects against these outcomes, this suggests the presence of residual confounding. Patients who have evidence of RZV during the six-month baseline period will be excluded from the negative control exposure analysis.

Similarly, potential negative control outcomes are outcomes that share the same sources of biases as the primary outcomes in our study population but are not causally-related to PCV13 vaccination. For example, immune status is an important predictor of pneumonia outcomes among PLWH, but we will be missing CD4 laboratory values for most of our study population. In order to detect potential residual confounding by lack of control for immune status, a potential negative control outcome could include a more common AIDS defining illness such as candidiasis. Again, if no residual confounding exists, PCV13 vaccination would have no effect on the occurrence of the negative control outcomes. However, if the results suggest that PCV13 vaccination prevents the negative control outcomes, residual confounding may exist.

If the negative control outcome analysis indicates residual confounding, the results of the main outcomes may be additionally reported after correcting for the bias [12].

## 5.8.9. Eligibility, Demographic, Clinical and Exposure Characteristics

The number and percentage of patients meeting the eligibility criteria will be reported in a subject evaluation table overall and by index calendar year.

Descriptive statistics will be used to summarize patient demographics and clinical characteristics of all PLWH using values at index date by vaccination status by the end of the baseline period. Overall SMDs will be presented before and after IPTW. SMDs at the end of each year since follow-up will also be tabulated.

Summaries of the overall follow-up time will be presented and calculated as time from index date to the earliest of death, end of health plan enrollment, or end of study period.

The number of patients who receive PCV13 by the end of the overall follow-up will be reported. Kaplan-Meier analysis will be used to summarize the percentage of persons who receive PCV13 by the end of each year of follow-up from index date. Patients will be censored at the earliest of the following: death, end of health plan enrollment, or end of study period.

The overall distributions of the IPT, IPC and IPT\*IPC weights will be summarized by vaccination status. To graphically assess the IPT weights over time a plot of the distributions of the log-transformed stabilized weights may also be presented at regular (e.g. six-monthly) intervals during the follow-up.

The above analysis will be repeated by the subgroups stated in Section 5.2.3.

## 5.8.10. Summaries of Study Outcomes

The number of patients with each study outcome will be presented by vaccination status at the time of infection (Table 5.2). Length of follow-up by PCV13 vaccination status will be presented by summarizing person-time before and after any PCV13 vaccine. Crude incidence rates and 95% CIs will be presented PCV13 vaccination status for each outcome for first episodes and again including recurrent episodes of the same type.

The above analysis will be repeated by the subgroups stated in Section .

#### 5.8.11. Analysis of Study Objectives

Crude HRs for PCV13 vaccination and the corresponding VE percentages will be presented together with 95% CIs for each study outcome overall and again during specific time periods (0-3, 3-5, 5-7 years). This will be done for first events and again including recurrent events. Analysis will be repeated using Cox-MSM after applying IPT and the IPT\*IPC weights.

The above analysis will be repeated by the subgroups stated in Section .

## 5.8.12. Analysis of Negative Control Outcomes and Exposure

The number of patients with the negative control outcome(s) will be presented by PCV13 vaccination status at the time of occurrence. Crude incidence rates and 95% CIs will be presented by PCV13 status for first and recurrent (separated by at least 90 days) episodes. Unadjusted and Cox-MSM will be used to obtain crude and weighted VE estimates and 95% CIs of PCV13 on candidiasis.

The number of patients who receive at least one dose of RZV by the end of the overall follow-up will be reported. Patients will be considered vaccinated with RZV 14 days after their vaccination date. Unadjusted and Cox-MSM will be used to obtain crude and weighted VE estimates and 95% CIs of RZV on each of the study outcomes of interest. Cox-MSM will additionally adjust for the main exposure of PCV13 as a time-varying covariate. Patients who have evidence of RZV before the six-month baseline period will be excluded from the negative control exposure analysis.

Weighted 95% CIs for the VEs that exclude 0% would suggest the presence of residual confounding in the weighted models between PCV13 and the study outcomes. If so, the results for the main outcomes may be corrected for bias identified from the negative control outcome.

## 6. REFERENCES

- Kobayashi, M., et al., Impact of 13-Valent Pneumococcal Conjugate Vaccine on Invasive Pneumococcal Disease Among Adults With HIV-United States, 2008-2018. J Acquir Immune Defic Syndr, 2022. 90(1): p. 6-14.
- Gierke, R. Current Epidemiology of Pneumococcal Disease, United States-2019 updates. June 25, 2021; Available from: https://www.cdc.gov/vaccines/acip/meetings/downloads/slides-2021-06/02-Pneumococcal-Gierke-508.pdf.
- Leidner, A. Summary of three economic models assessing pneumococcal vaccines in US adults. September 29, 2021; Available from: https://www.cdc.gov/vaccines/acip/meetings/downloads/slides-2021-09-29/02-Pneumococcal-Leidner-508.pdf.
- Hsiao, A., et al., Incidence and Estimated Vaccine Effectiveness Against
  Hospitalizations for All-Cause Pneumonia Among Older US Adults Who Were
  Vaccinated and Not Vaccinated With 13-Valent Pneumococcal Conjugate Vaccine.
  JAMA Netw Open, 2022. 5(3): p. e221111.
- 5. Austin, P.C., Generating survival times to simulate Cox proportional hazards models with time-varying covariates. Stat Med, 2012. 31(29): p. 3946-58.
- CDC's Social Vulnerability Index (SVI). November 30, 2022]; Available from: https://www.atsdr.cdc.gov/placeandhealth/svi/index.html.
- Hyer, J.M., et al., High Social Vulnerability and "Textbook Outcomes" after Cancer Operation. J Am Coll Surg, 2021. 232(4): p. 351-359.
- 8. de Oliveira Costa, J., et al., Assessing the impact of implementing multiple adherence measures to antiretroviral therapy from dispensing data: a short report. AIDS Care, 2022: p. 1-6.
- Cole, S.R. and M.A. Hernan, Constructing inverse probability weights for marginal structural models. Am J Epidemiol, 2008. 168(6): p. 656-64.
- van der Wal, W.M. and R.B. Geskus, ipw: An R Package for Inverse Probability Weighting. Journal of Statistical Software, 2011. 43(13): p. 1 - 23.
- Andersen, P.K. and R.D. Gill, Cox's Regression Model for Counting Processes: A Large Sample Study. The Annals of Statistics, 1982. 10(4): p. 1100-1120, 21.
- Tchetgen Tchetgen, E.J.S., Tamar; Richardson, David, Negative Outcome Control for Unobserved Confounding Under a Cox Proportional Hazards Model. Harvard University Biostatistics Working Paper Series. Working Paper 192., July 2015.

## 7. APPENDICES

## 7.1. Appendix A: Table shells

The list of planned outputs and table shells will be presented in a separate document.

# 7.2. Appendix B: R Example Code

# 7.2.1. Example Data Formats for First Event and Recurrent Events

Example dataset for time to first outcome:

| ptid | tstart | tstop | pcv13 | ipd | x1 | <b>x</b> 2 | xt1 | xt2 | censor | endfu |
|---|---|---|---|---|---|---|---|---|---|---|
| 1001 | -1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 87 |
| 1001 | 0 | 30 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 87 |
| 1001 | 30 | 60 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 87 |
| 1001 | 60 | 87 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 87 |
| 1002 | -1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 45 |
| 1002 | 0 | 30 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 45 |
| 1002 | 30 | 45 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 45 |

Example dataset including any subsequent outcomes:

| ptid | tstart | tstop | pcv13 | ipd | x1 | <b>x</b> 2 | xt1 | xt2 | censor | endfu2 |
|---|---|---|---|---|---|---|---|---|---|---|
| 1001 | -1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 87 |
| 1001 | 0 | 30 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 87 |
| 1001 | 30 | 60 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 87 |
| 1001 | 60 | 87 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 87 |
| 1002 | -1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 106 |
| 1002 | 0 | 30 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 106 |
| 1002 | 30 | 45 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 106 |
| 1002 | 45 | 60 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 106 |
| 1002 | 60 | 84 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 106 |
| 1002 | 84 | 90 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 106 |
| 1002 | 90 | 106 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 106 |

## Where:

- ptid: patient identifier
- tstart: first day of interval. -1 represents baseline period
- tstop: last day of interval
- pcv13: binary indicator for time-varying PCV13 vaccination status (exposure)
- ipd: binary indicator for IPD event (outcome)
- x1, x2, ..., xn: time-fixed confounders
- xt1, xt2, ..., xtn: time-varying confounders
- censor: binary indicator for censoring event

- endfu: last day of follow-up up to any first event
- endfu2: last day of follow-up

SAP version 1.3,07 December 2023

For binary variables, 1 indicates Yes, 0 indicates No. Note, all variables in dataset must be numeric for the *ipwtm* function.

# 7.2.2. Code for Generating IPTW and IPCW

```
library(ipw)
iptw <- ipwtm(exposure = pcv13, family = "survival",
numerator = \sim x1 + x2 + \dots + xn, denominator = \sim x1 + x2 + \dots + xn + xt1 + xt2 + \dots + xtn,
id = ptid, tstart = tstart, timevar = tstop, type = "first",
data = ipdfirst
ipcw <- ipwtm(exposure = censor, family = "survival",
numerator = \sim x1 + x2 + \dots + xn, denominator = \sim x1 + x2 + \dots + xn + xt1 + xt2 + \dots + xtn,
        id = patient, tstart = tstart, timevar = tstop, type = "cens",
         data = ipdfirst)
iptw.stab<-iptw$ipw.weights
ipcw.stab<-ipcw$ipw.weights
ipdfirst<-cbind(ipdfirst, iptw.stab, ipcw.stab)
ipdfirst$comb.weights<- ipdfirst$ iptw.stab*ipdfirst$ ipcw.stab
#Plot of stabilized weights during follow-up in unvaccinated
ipwplot(weights = subset(ipdfirst$iptw, ipdifrst$pcv13==0),
       subset(timevar = ipdfirst$tstop, ipdifrst$pcv13==0),
       binwidth = 183, ylim = c(-1.5, 1.5), main = "Stabilized weights",
       xlab = "Years Since Index", ylab = "Logarithm of Stabilized IPTW",
xaxt = "n", yaxt = "n"
axis(side = 1, at = seq(0, 15, 1),
                                   labels = as.character(seq(0,15,1)*0.5))
axis(side = 2, at = c(-1.5, -1, -0.5, 0, 0.5, 1, 1.5),
   labels = as.character(c(-1.5, -1, -0.5, 0, 0.5, 1, 1.5))
7.2.3. Code for Incidence Rates
#First events
ipdfirst$py <-ifelse(ipdfirst$tstart>=0,
             (ipdfirst$tstop - ipdfirst$tstart)/365.25,0)
ipdfirst$lnpy <-ifelse(ipdfirst$tstart>=0,log(ipdfirst$py),0)
#Rate in unvaccinated
fit erate unvac <- glm(event ~ pcv13 + offset(lnpy), family=poisson(link="log"),
```

subset(ipdfirst[ipdfirst\$tstart>=0, ]))

summary(fit erate unvac) exp(coef(fit erate unvac)[1])

```
exp(confint(fit erate unvac))
#Rate in vaccinated (where pcv13 is factor)
fit erate vac <- glm(event ~ relevel(pcv13, ref="1") + offset(lnpy),
   family= poisson(link="log"), subset(ipdfirst[ipdfirst$tstart>=0, ]))
summary(fit erate vac)
exp(coef(fit erate vac)[1])
exp(confint(fit_erate_vac))
#Recurrent events
library("sandwich")
library("lmtest")
#Rate in unvaccinated
fit erate rec unvac <- glm(event ~ pcv13 + offset(lnpy), family=poisson(link="log"),
          subset(ipdrec[ipdrec$tstart>=0, ]))
fit_clust_rec_unvac <-coeftest(fit_erate_rec_unvac, vcov. = vcovCL(fit_erate_rec_unvac,
                            cluster = ipdrec$patid, type = "HC0"))
fit clust rec unvac
exp(coef(fit clust rec unvac)[1])
exp(confint(fit clust rec unvac))
#Rate in vaccinated (where pcv13 is factor)
fit erate rec vac <- glm(event ~ relevel(pcv13, ref="1") + offset(lnpy),
    family=poisson(link="log"), subset(ipdrec[ipdrec$tstart>=0, ]))
fit clust rec vac <-coeftest(fit erate rec vac, vcov. = vcovCL(fit erate rec vac,
                            cluster = ipdrec$patid, type = "HC0"))
fit clust rec vac
exp(coef(fit clust rec vac)[1])
exp(confint(fit clust rec vac))
7.2.4. Code for Standardized Differences
library(cobalt)
smdDataY1<-subset(ipdfirst[ipdfirst$tstart==360 &
                (ipdfirst$tstart < ipdfirst$pcv13date14 | is.na(ipdfirst$ pcv13date14)),])
#Where pcv13date14 is 14 days after the PCV13 vaccination date
covs \le subset(smdDataY1, select = c(x1, x2, ...))
#Before IPTW
smdsUn<-bal.tab(covs, treat = smdDataY1$pcv13, continuous = "std",</pre>
        binary = "std", s.d.denom = "pooled")
x1SmdUn<-smdsUn$Balance[1,2]
x2SmdUn<-smdsUn$Balance[2,2]
#After IPTW
smdsWt<-bal.tab(covs, treat = smdDataY1$pcv13, continuous = "std",</pre>
```

publish(iptw.cox.p)

```
binary = "std", s.d.denom = "pooled", weights=smdDataY1$iptw.stab)
x1SmdWt<-smdsWt$Balance[1,3]
x2SmdWt<-smdsWt$Balance[2,3]
7.2.5. Code for Cox Models
#Code is the same for first event and recurrent events (Andersen-Gill) models
#Crude overall
library(survival)
crude.cox<-coxph(Surv(tstart, tstop, ipd) ~ pcv13 + cluster(ptid), data = ipdfirst)
#IPT weighted overall
iptw.cox<-coxph(Surv(tstart, tstop, ipd) \sim pcv13 + x1 + x2 + cluster(ptid),
       data = ipdfirst), weights = iptw.stab
# Schoenfeld residuals
plot(cox.zph(iptw.cox)[1])
#Piecewise IPT weighted
library(Publish)
ipdfirst$timestrata<-ifelse(ipdfirst$tstart<1080,"0-3",
       ifelse(ipdfirst$tstart<1800,"3-5", ifelse(ipdfirst$tstart<2550,"5-7","7+")))
iptw.cox.p<-coxph(Surv(tstart, tstop, ipd) \sim pcv13*strata(timestrata) + x1 + x2 +
       cluster(ptid), data = ipdfirst, weights = iptw.stab)
summary(iptw.cox.p)
```

# 7.3. Appendix C: Diagnosis and Procedure Codes Used in the Study

Table 7.1 Diagnosis Codes for Identifying HIV Infection

| Code | Type | Description |
|------|-----------|--------------------------|
| 042 | ICD-9-CM | HIV-1 infection |
| V08 | ICD-9-CM | Asymptomatic HIV disease |
| B20 | ICD-10-CM | HIV-1 infection |
| Z21 | ICD-10-CM | Asymptomatic HIV disease |

Table 7.2 National Drug Codes for Identifying HIV Antiretrovirals (see Excel)

Table 7.3 NDC and CPT Codes for Identifying PCV13 Vaccination

| Code | Type | Description |
|-------------|------|------------------------------------------|
| 50090194409 | NDC | 13-valent pneumococcal conjugate vaccine |
| 54569661300 | NDC | 13-valent pneumococcal conjugate vaccine |
| 50090194400 | NDC | 13-valent pneumococcal conjugate vaccine |
| 00005197105 | NDC | 13-valent pneumococcal conjugate vaccine |
| 00005197104 | NDC | 13-valent pneumococcal conjugate vaccine |
| 00005197102 | NDC | 13-valent pneumococcal conjugate vaccine |
| 00005197101 | NDC | 13-valent pneumococcal conjugate vaccine |
| 90670 | СРТ | 13-valent pneumococcal conjugate vaccine |

Table 7.4 Diagnosis Codes for Identifying Invasive Pneumococcal Disease, All-Cause Pneumonia, and Pneumococcal Pneumonia

| | ICD-9-CM | | | ICD-10-CM |
|---|---|---|---|---|
| Condition | Codes | Description | Codes | Description |
| IPD | | | | |
| | 790.7 + 041.2<br>771.83 +<br>041.2 | Bacteremia + pneumococcus | R78.81 + B95.3 | Bacteremia + Streptococcus pneumoniae as the cause of diseases classified elsewhere (Streptococcus pneumoniae) |
| Bacteremia | 038.2 | Pneumococcal septicemia | A40.3 | Sepsis due to Streptococcus pneumoniae |
| | 038.9 + 041.2 | 038.9 + 041.2 Unspecified septicemia + pneumococcus A41.9 | | Sepsis, unspecified organism + Streptococcus pneumoniae |
| | 320.1 | Pneumococcal meningitis | G00.1 | Pneumococcal meningitis |
| Meningitis | 320.9 + 041.2 | Meningitis due to unspecified<br>bacterium + pneumococcus | G00.9 + B95.3<br>G04.2 + B95.3 | Bacterial meningitis, unspecified + Streptococcus pneumoniae<br>Bacterial meningoencephalitis and meningomyelitis, not elsewhere classified +<br>Streptococcus pneumoniae |
| | 322.9 + 041.2 | Meningitis, unspecified + pneumococcus | G03.9 + B95.3 | Meningitis, unspecified + Streptococcus pneumoniae |
| | 421.x + 041.2 | | Endo | ocarditis + pneumococcus |
| Other | 421 + 041.2 | Acute and subacute bacterial<br>endocarditis + pneumococcus | I33.0 + B95.3 | Acute and subacute infective endocarditis + Streptococcus pneumoniae |
| | 421.1 + 041.2 | Acute and subacute infective<br>endocarditis in diseases<br>classified elsewhere +<br>pneumococcus | I39 + B95.3 | Endocarditis and heart valve disorders in diseases classified elsewhere +<br>Streptococcus pneumoniae |

| 421.9 + 0 | Acute endocarditis,<br>unspecified + pneumococcus | I33.9 + B95.3 | Acute and subacute endocarditis, unspecified + Streptococcus pneumoniae |
|---|---|---|---|
| 711.0 + 0 | Septic arthritis + pneumococcus | M00.00 + B95.3<br>M00.20 + B95.3<br>M00.80 + B95.3<br>M00.9 + B95.3<br>M00.10 + B95.3 | Staphylococcal arthritis, unspecified joint + Streptococcus pneumoniae Other streptococcal arthritis, unspecified joint + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified joint + Streptococcus pneumoniae Pyogenic arthritis, unspecified + Streptococcus pneumoniae Pneumococcal arthritis, unspecified joint + Streptococcus pneumoniae |
| 711.01<br>041.1 | - ) - 8 , | M00.011 + B95.3<br>M00.012 + B95.3<br>M00.019 + B95.3<br>M00.211 + B95.3<br>M00.212 + B95.3<br>M00.219 + B95.3<br>M00.811 + B95.3<br>M00.812 + B95.3<br>M00.819 + B95.3<br>M00.119 + B95.3<br>M00.111 + B95.3<br>M00.112 + B95.3 | Staphylococcal arthritis, right shoulder + Streptococcus pneumoniae Staphylococcal arthritis, left shoulder + Streptococcus pneumoniae Staphylococcal arthritis, unspecified shoulder + Streptococcus pneumoniae Other streptococcal arthritis, left shoulder + Streptococcus pneumoniae Other streptococcal arthritis, left shoulder + Streptococcus pneumoniae Other streptococcal arthritis, unspecified shoulder + Streptococcus pneumoniae Arthritis due to other bacteria, right shoulder + Streptococcus pneumoniae Arthritis due to other bacteria, left shoulder + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified shoulder + Streptococcus pneumoniae Pneumococcal arthritis, unspecified shoulder + Streptococcus pneumoniae Pneumococcal arthritis, right shoulder + Streptococcus pneumoniae Pneumococcal arthritis, left shoulder + Streptococcus pneumoniae |
| 711.02<br>041.1 | - ) - B , -FF | M00.021 + B95.3<br>M00.022 + B95.3<br>M00.029 + B95.3<br>M00.221 + B95.3<br>M00.222 + B95.3<br>M00.229 + B95.3<br>M00.821 + B95.3<br>M00.822 + B95.3<br>M00.829 + B95.3<br>M00.129 + B95.3<br>M00.129 + B95.3 | Staphylococcal arthritis, right elbow + Streptococcus pneumoniae Staphylococcal arthritis, left elbow + Streptococcus pneumoniae Staphylococcal arthritis, unspecified elbow + Streptococcus pneumoniae Other streptococcal arthritis, right elbow + Streptococcus pneumoniae Other streptococcal arthritis, left elbow + Streptococcus pneumoniae Other streptococcal arthritis, unspecified elbow + Streptococcus pneumoniae Arthritis due to other bacteria, right elbow + Streptococcus pneumoniae Arthritis due to other bacteria, left elbow + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified elbow + Streptococcus pneumoniae Pneumococcal arthritis, unspecified elbow + Streptococcus pneumoniae Pneumococcal arthritis, right elbow + Streptococcus pneumoniae Pneumococcal arthritis, left elbow + Streptococcus pneumoniae |
| 711.03<br>041. | - j -g, | M00.031 + B95.3<br>M00.032 + B95.3<br>M00.039 + B95.3<br>M00.231 + B95.3 | Staphylococcal arthritis, right wrist + Streptococcus pneumoniae Staphylococcal arthritis, left wrist + Streptococcus pneumoniae Staphylococcal arthritis, unspecified wrist + Streptococcus pneumoniae Other streptococcal arthritis, right wrist + Streptococcus pneumoniae |

| 711.04 +<br>041.2 | Pyogenic arthritis, hand + pneumococcus | M00.239 + B95.3<br>M00.831 + B95.3<br>M00.832 + B95.3<br>M00.839 + B95.3<br>M00.139 + B95.3<br>M00.131 + B95.3<br>M00.132 + B95.3<br>M00.042 + B95.3<br>M00.042 + B95.3<br>M00.241 + B95.3<br>M00.242 + B95.3<br>M00.249 + B95.3<br>M00.841 + B95.3<br>M00.842 + B95.3<br>M00.842 + B95.3<br>M00.149 + B95.3<br>M00.149 + B95.3<br>M00.149 + B95.3<br>M00.149 + B95.3 | Other streptococcal arthritis, unspecified wrist + Streptococcus pneumoniae Arthritis due to other bacteria, left wrist + Streptococcus pneumoniae Arthritis due to other bacteria, left wrist + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified wrist + Streptococcus pneumoniae Pneumococcal arthritis, unspecified wrist + Streptococcus pneumoniae Pneumococcal arthritis, right wrist + Streptococcus pneumoniae Pneumococcal arthritis, left wrist + Streptococcus pneumoniae Staphylococcal arthritis, left hand + Streptococcus pneumoniae Staphylococcal arthritis, unspecified hand + Streptococcus pneumoniae Other streptococcal arthritis, left hand + Streptococcus pneumoniae Other streptococcal arthritis, left hand + Streptococcus pneumoniae Other streptococcal arthritis, unspecified hand + Streptococcus pneumoniae Arthritis due to other bacteria, right hand + Streptococcus pneumoniae Arthritis due to other bacteria, left hand + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified hand + Streptococcus pneumoniae Pneumococcal arthritis, unspecified hand + Streptococcus pneumoniae Pneumococcal arthritis, right hand + Streptococcus pneumoniae Pneumococcal arthritis, left hand + Streptococcus pneumoniae Pneumococcal arthritis, left hand + Streptococcus pneumoniae Pneumococcal arthritis, left hand + Streptococcus pneumoniae |
|---|---|---|---|
| 711.05 +<br>041.2 | Pyogenic arthritis, pelvic<br>region and thigh +<br>pneumococcus | M00.051 + B95.3<br>M00.052 + B95.3<br>M00.059 + B95.3<br>M00.251 + B95.3<br>M00.252 + B95.3<br>M00.259 + B95.3<br>M00.851 + B95.3<br>M00.852 + B95.3<br>M00.859 + B95.3<br>M00.159 + B95.3<br>M00.151 + B95.3<br>M00.152 + B95.3 | Staphylococcal arthritis, right hip + Streptococcus pneumoniae Staphylococcal arthritis, left hip + Streptococcus pneumoniae Staphylococcal arthritis, unspecified hip + Streptococcus pneumoniae Other streptococcal arthritis, right hip + Streptococcus pneumoniae Other streptococcal arthritis, left hip + Streptococcus pneumoniae Other streptococcal arthritis, unspecified hip + Streptococcus pneumoniae Arthritis due to other bacteria, right hip + Streptococcus pneumoniae Arthritis due to other bacteria, left hip + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified hip + Streptococcus pneumoniae Pneumococcal arthritis, unspecified hip + Streptococcus pneumoniae Pneumococcal arthritis, right hip + Streptococcus pneumoniae Pneumococcal arthritis, left hip + Streptococcus pneumoniae |

| 711.06 +<br>041.2 | Pyogenic arthritis, lower leg + pneumococcus | M00.061 + B95.3<br>M00.062 + B95.3<br>M00.069 + B95.3<br>M00.261 + B95.3<br>M00.262 + B95.3<br>M00.269 + B95.3<br>M00.861 + B95.3<br>M00.862 + B95.3<br>M00.869 + B95.3<br>M00.169 + B95.3<br>M00.161 + B95.3<br>M00.162 + B95.3 | Staphylococcal arthritis, right knee + Streptococcus pneumoniae Staphylococcal arthritis, left knee + Streptococcus pneumoniae Staphylococcal arthritis, unspecified knee + Streptococcus pneumoniae Other streptococcal arthritis, right knee + Streptococcus pneumoniae Other streptococcal arthritis, left knee + Streptococcus pneumoniae Other streptococcal arthritis, unspecified knee + Streptococcus pneumoniae Arthritis due to other bacteria, right knee + Streptococcus pneumoniae Arthritis due to other bacteria, left knee + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified knee + Streptococcus pneumoniae Pneumococcal arthritis, unspecified knee + Streptococcus pneumoniae Pneumococcal arthritis, right knee + Streptococcus pneumoniae Pneumococcal arthritis, left knee + Streptococcus pneumoniae |
|---|---|---|---|
| 711.07 +<br>041.2 | Pyogenic arthritis, ankle and<br>foot + pneumococcus | M00.071 + B95.3<br>M00.072 + B95.3<br>M00.079 + B95.3<br>M00.271 + B95.3<br>M00.272 + B95.3<br>M00.279 + B95.3<br>M00.871 + B95.3<br>M00.872 + B95.3<br>M00.879 + B95.3<br>M00.179 + B95.3<br>M00.179 + B95.3<br>M00.171 + B95.3 | Staphylococcal arthritis, right ankle and foot + Streptococcus pneumoniae Staphylococcal arthritis, left ankle and foot + Streptococcus pneumoniae Staphylococcal arthritis, unspecified ankle and foot + Streptococcus pneumoniae Other streptococcal arthritis, right ankle and foot + Streptococcus pneumoniae Other streptococcal arthritis, left ankle and foot + Streptococcus pneumoniae Other streptococcal arthritis, unspecified ankle and foot + Streptococcus pneumoniae Arthritis due to other bacteria, right ankle and foot + Streptococcus pneumoniae Arthritis due to other bacteria, left ankle and foot + Streptococcus pneumoniae Arthritis due to other bacteria, unspecified ankle and foot + Streptococcus pneumoniae Pneumococcal arthritis, unspecified ankle and foot + Streptococcus pneumoniae Pneumococcal arthritis, right ankle and foot + Streptococcus pneumoniae Pneumococcal arthritis, left ankle and foot + Streptococcus pneumoniae |
| 711.08 +<br>041.2 | Pyogenic arthritis, other<br>specified sites +<br>pneumococcus | M00.08 + B95.3<br>M00.28 + B95.3<br>M00.88 + B95.3<br>M00.9+ B95.3<br>M00.18 + B95.3 | Staphylococcal arthritis, vertebrae + Streptococcus pneumoniae Other streptococcal arthritis, vertebrae + Streptococcus pneumoniae Arthritis due to other bacteria, vertebrae + Streptococcus pneumoniae Pyogenic arthritis, unspecified + Streptococcus pneumoniae Pneumococcal arthritis, vertebrae + Streptococcus pneumoniae |
| 711.09 +<br>041.2 | Pyogenic arthritis, multiple<br>sites + pneumococcus | M00.09 + B95.3<br>M00.29 + B95.3<br>M00.89 + B95.3<br>M00.19 + B95.3 | Staphylococcal polyarthritis + Streptococcus pneumoniae Other streptococcal polyarthritis + Streptococcus pneumoniae Polyarthritis due to other bacteria + Streptococcus pneumoniae Pneumococcal polyarthritis + Streptococcus pneumoniae |

| 730.0x +<br>041.2<br>730.2x +<br>041.2 | | Oste | omyelitis + pneumococcus |
|---|---|---|---|
| 730.00 +<br>041.2 | Acute osteomyelitis, site<br>unspecified + pneumococcus | M86.00 + B95.3<br>M86.10 + B95.3<br>M86.20 + B95.3 | Acute hematogenous osteomyelitis, unspecified site + Streptococcus pneumoniae Other acute osteomyelitis, unspecified site + Streptococcus pneumoniae Subacute osteomyelitis, unspecified site + Streptococcus pneumoniae |
| 730.01 +<br>041.2 | Acute osteomyelitis, shoulder region + pneumococcus | M86.011 + B95.3<br>M86.012 + B95.3<br>M86.019 + B95.3<br>M86.111 + B95.3<br>M86.112 + B95.3<br>M86.119 + B95.3<br>M86.211 + B95.3<br>M86.212 + B95.3<br>M86.219 + B95.3 | Acute hematogenous osteomyelitis, right shoulder + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left shoulder + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified shoulder + Streptococcus pneumoniae Other acute osteomyelitis, right shoulder + Streptococcus pneumoniae Other acute osteomyelitis, left shoulder + Streptococcus pneumoniae Other acute osteomyelitis, unspecified shoulder + Streptococcus pneumoniae Subacute osteomyelitis, right shoulder + Streptococcus pneumoniae Subacute osteomyelitis, left shoulder + Streptococcus pneumoniae Subacute osteomyelitis, unspecified shoulder + Streptococcus pneumoniae |
| 730.02 +<br>041.2 | Acute osteomyelitis, upper<br>arm + pneumococcus | M86.021 + B95.3<br>M86.022 + B95.3<br>M86.029 + B95.3<br>M86.121 + B95.3<br>M86.122 + B95.3<br>M86.129 + B95.3<br>M86.221 + B95.3<br>M86.222 + B95.3<br>M86.222 + B95.3 | Acute hematogenous osteomyelitis, right humerus + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left humerus + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified humerus + Streptococcus pneumoniae Other acute osteomyelitis, right humerus + Streptococcus pneumoniae Other acute osteomyelitis, left humerus + Streptococcus pneumoniae Other acute osteomyelitis, unspecified humerus + Streptococcus pneumoniae Subacute osteomyelitis, right humerus + Streptococcus pneumoniae Subacute osteomyelitis, left humerus + Streptococcus pneumoniae Subacute osteomyelitis, unspecified humerus + Streptococcus pneumoniae |
| 730.03 +<br>041.2 | Acute osteomyelitis, forearm | M86.031 + B95.3<br>M86.032 + B95.3<br>M86.039 + B95.3<br>M86.131 + B95.3<br>M86.132 + B95.3<br>M86.139 + B95.3<br>M86.231 + B95.3 | Acute hematogenous osteomyelitis, right radius and ulna + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left radius and ulna + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified radius and ulna + Streptococcus pneumoniae Other acute osteomyelitis, right radius and ulna + Streptococcus pneumoniae Other acute osteomyelitis, left radius and ulna + Streptococcus pneumoniae |

| | | | M86.232 + B95.3<br>M86.239 + B95.3 | Other acute osteomyelitis, unspecified radius and ulna + Streptococcus pneumoniae Subacute osteomyelitis, right radius and ulna + Streptococcus pneumoniae Subacute osteomyelitis, left radius and ulna + Streptococcus pneumoniae Subacute osteomyelitis, unspecified radius and ulna + Streptococcus pneumoniae |
|--|---|---|---|---|
| | 730.04 +<br>041.2 | Acute osteomyelitis, hand + pneumococcus | M86.041 + B95.3<br>M86.042 + B95.3<br>M86.049 + B95.3<br>M86.141 + B95.3<br>M86.142 + B95.3<br>M86.149 + B95.3<br>M86.241 + B95.3<br>M86.242 + B95.3<br>M86.249 + B95.3 | Acute hematogenous osteomyelitis, right hand + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left hand + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified hand + Streptococcus pneumoniae Other acute osteomyelitis, right hand + Streptococcus pneumoniae Other acute osteomyelitis, left hand + Streptococcus pneumoniae Other acute osteomyelitis, unspecified hand + Streptococcus pneumoniae Subacute osteomyelitis, right hand + Streptococcus pneumoniae Subacute osteomyelitis, left hand + Streptococcus pneumoniae Subacute osteomyelitis, unspecified hand + Streptococcus pneumoniae |
| | 730.05 +<br>041.2 | Acute osteomyelitis, pelvic<br>region and thigh +<br>pneumococcus | M86.051 + B95.3<br>M86.052 + B95.3<br>M86.059 + B95.3<br>M86.151 + B95.3<br>M86.152 + B95.3<br>M86.159 + B95.3<br>M86.251 + B95.3<br>M86.252 + B95.3<br>M86.259 + B95.3 | Acute hematogenous osteomyelitis, right femur + Streptococcus pneumonia Acute hematogenous osteomyelitis, left femur + Streptococcus pneumonia Acute hematogenous osteomyelitis, unspecified femur + Streptococcus pneumonia Other acute osteomyelitis, right femur + Streptococcus pneumonia Other acute osteomyelitis, left femur + Streptococcus pneumonia Other acute osteomyelitis, unspecified femur + Streptococcus pneumonia Subacute osteomyelitis, right femur + Streptococcus pneumoniae Subacute osteomyelitis, left femur + Streptococcus pneumoniae Subacute osteomyelitis, unspecified femur + Streptococcus pneumoniae |
| | 730.06 +<br>041.2 | Acute osteomyelitis, lower leg<br>+ pneumococcus | M86.061 + B95.3<br>M86.062 + B95.3<br>M86.069 + B95.3<br>M86.161 + B95.3<br>M86.162 + B95.3<br>M86.169 + B95.3<br>M86.261 + B95.3<br>M86.262 + B95.3<br>M86.269 + B95.3 | Acute hematogenous osteomyelitis, right tibia and fibula + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left tibia and fibula + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified tibia and fibula + Streptococcus pneumoniae Other acute osteomyelitis, right tibia and fibula + Streptococcus pneumoniae Other acute osteomyelitis, left tibia and fibula + Streptococcus pneumoniae Other acute osteomyelitis, unspecified tibia and fibula + Streptococcus pneumoniae Subacute osteomyelitis, right tibia and fibula + Streptococcus pneumoniae Subacute osteomyelitis, left tibia and fibula + Streptococcus pneumoniae Subacute osteomyelitis, unspecified tibia and fibula + Streptococcus pneumoniae |
| 730.07 +<br>041.2 | Acute osteomyelitis, ankle and foot + pneumococcus | M86.071 + B95.3<br>M86.072 + B95.3<br>M86.079 + B95.3<br>M86.171 + B95.3<br>M86.172 + B95.3<br>M86.179 + B95.3<br>M86.271 + B95.3<br>M86.272 + B95.3<br>M86.279 + B95.3 | Acute hematogenous osteomyelitis, right ankle and foot + Streptococcus pneumoniae Acute hematogenous osteomyelitis, left ankle and foot + Streptococcus pneumoniae Acute hematogenous osteomyelitis, unspecified ankle and foot + Streptococcus pneumoniae Other acute osteomyelitis, right ankle and foot + Streptococcus pneumoniae Other acute osteomyelitis, left ankle and foot + Streptococcus pneumoniae Other acute osteomyelitis, unspecified ankle and foot + Streptococcus pneumoniae Subacute osteomyelitis, right ankle and foot + Streptococcus pneumoniae Subacute osteomyelitis, unspecified ankle and foot + Streptococcus pneumoniae Subacute osteomyelitis, unspecified ankle and foot + Streptococcus pneumoniae |
|---|---|---|---|
| 730.08 +<br>041.2 | Acute osteomyelitis, other<br>specified sites +<br>pneumococcus | M86.08 + B95.3<br>M86.18 + B95.3<br>M86.28 + B95.3 | Acute hematogenous osteomyelitis, other sites + Streptococcus pneumoniae Other acute osteomyelitis, other site + Streptococcus pneumoniae Subacute osteomyelitis, other site + Streptococcus pneumoniae |
| 730.09 +<br>041.2 | Acute osteomyelitis, multiple sites<br>+ pneumococcus | M86.09 + B95.3<br>M86.19 + B95.3<br>M86.29 + B95.3 | Acute hematogenous osteomyelitis, multiple sites + Streptococcus pneumoniae Other acute osteomyelitis, multiple sites + Streptococcus pneumoniae Subacute osteomyelitis, multiple sites + Streptococcus pneumoniae |
| 730.2 + 041.2<br>730.21 +<br>041.2<br>730.22 +<br>041.2<br>730.23 +<br>041.2<br>730.24 +<br>041.2<br>730.25 +<br>041.2<br>730.26 +<br>041.2<br>730.27 +<br>041.2<br>730.29 +<br>041.2 | Unspecified osteomyelitis, site unspecified + pneumococcus Unspecified osteomyelitis, shoulder region + pneumococcus Unspecified osteomyelitis, upper arm + pneumococcus Unspecified osteomyelitis, forearm + pneumococcus Unspecified osteomyelitis, hand + pneumococcus Unspecified osteomyelitis, pelvic region and thigh + pneumococcus Unspecified osteomyelitis, lower leg + pneumococcus Unspecified osteomyelitis, ankle and foot + pneumococcus Unspecified osteomyelitis, multiple sites + pneumococcus | M86.9 + B95.3 | Osteomyelitis, unspecified + Streptococcus pneumoniae |

| | 730.28 +<br>041.2 | Unspecified osteomyelitis,<br>other specified sites +<br>pneumococcus | M46.20 + B95.3<br>M46.21 + B95.3<br>M46.22 + B95.3<br>M46.23 + B95.3<br>M46.24 + B95.3<br>M46.25 + B95.3<br>M46.26 + B95.3<br>M46.27 + B95.3<br>M46.28 + B95.3 | Osteomyelitis of vertebra, site unspecified + Streptococcus pneumoniae Osteomyelitis of vertebra, occipito-atlanto-axial region + Streptococcus pneumoniae Osteomyelitis of vertebra, cervical region + Streptococcus pneumoniae Osteomyelitis of vertebra, cervicothoracic region + Streptococcus pneumoniae Osteomyelitis of vertebra, thoracic region + Streptococcus pneumoniae Osteomyelitis of vertebra, thoracolumbar region + Streptococcus pneumoniae Osteomyelitis of vertebra, lumbar region + Streptococcus pneumoniae Osteomyelitis of vertebra, lumbosacral region + Streptococcus pneumoniae Osteomyelitis of vertebra, sacral and sacrococcygeal region + Streptococcus pneumoniae |
|---|---|---|---|---|
| Pneumonia | | | | |
| | 480-486<br>487.0 | | Viral, ba | cterial, unspecified pneumonia |
| | 480 | Pneumonia due to adenovirus | J12.0 | Adenoviral pneumonia |
| | 480.1 | Pneumonia due to respiratory<br>syncytial virus | J12.1 | Respiratory syncytial virus pneumonia |
| | 480.2 | Pneumonia due to<br>parainfluenza virus | J12.2 | Parainfluenza virus pneumonia |
| All-Cause | 480.3 | Pneumonia due to SARS- | J12.81 | Pneumonia due to SARS-associated coronavirus |
| | 400.3 | associated coronavirus | J12.82 | Pneumonia due to coronavirus disease 2019 |
| | 480.8 | Pneumonia due to other virus<br>not elsewhere classified | J12.3<br>J12.89 | Human metapneumovirus pneumonia<br>Other viral pneumonia |
| | 480.9 | Viral pneumonia, unspecified | J12.9 | Viral pneumonia, unspecified |
| | 481 | Pneumococcal pneumonia<br>[Streptococcus pneumoniae<br>pneumonia] | J18.1<br>J13 | Lobar pneumonia, unspecified organism Pneumonia due to Streptococcus pneumoniae |

| 482 | Pneumonia due to Klebsiella<br>pneumoniae | J15.0 | Pneumonia due to Klebsiella pneumoniae |
|---|---|---|---|
| 482.1 | Pneumonia due to<br>Pseudomonas | J15.1 | Pneumonia due to Pseudomonas |
| 482.2 | Pneumonia due to Hemophilus<br>influenzae [H. influenzae] | J14 | Pneumonia due to Hemophilus influenzae |
| 482.3 | Pneumonia due to<br>Streptococcus, unspecified | J15.4 | Pneumonia due to other streptococci |
| 482.31 | Pneumonia due to<br>Streptococcus, group A | J15.4 | Pneumonia due to other streptococci |
| 482.32 | Pneumonia due to<br>Streptococcus, group B | J15.3 | Pneumonia due to streptococcus, group B |
| 482.39 | Pneumonia due to other<br>Streptococcus | J15.4 | Pneumonia due to other streptococci |
| 482.4 | Pneumonia due to<br>Staphylococcus, unspecified | J15.20 | Pneumonia due to staphylococcus, unspecified |
| 482.41 | Methicillin susceptible<br>pneumonia due to<br>Staphylococcus aureus | J15.211 | Pneumonia due to Methicillin susceptible Staphylococcus aureus |
| 482.42 | Methicillin resistant<br>pneumonia due to<br>Staphylococcus aureus | J15.212 | Pneumonia due to Methicillin resistant Staphylococcus aureus |
| 482.49 | Other Staphylococcus<br>pneumonia | J15.29 | Pneumonia due to other staphylococcus |
| 482.81 | Pneumonia due to anaerobes | J15.8 | Pneumonia due to other specified bacteria |

| 482.82 | Pneumonia due to escherichia<br>coli [E. coli] | J15.5 | Pneumonia due to Escherichia coli |
|---|---|---|---|
| 482.83 | Pneumonia due to other gram-<br>negative bacteria | J15.6 | Pneumonia due to other aerobic Gram-negative bacteria |
| 482.84 | Pneumonia due to<br>Legionnaires' disease | A48.1 | Legionnaires' disease |
| 482.89 | Pneumonia due to other<br>specified bacteria | J15.8 | Pneumonia due to other specified bacteria |
| 482.9 | Bacterial pneumonia,<br>unspecified | J15.9 | Unspecified bacterial pneumonia |
| 483 | Pneumonia due to<br>mycoplasma pneumoniae | J15.7 | Pneumonia due to Mycoplasma pneumoniae |
| 483.1 | Pneumonia due to chlamydia | J16.0 | Chlamydial pneumonia |
| 483.8 | Pneumonia due to other<br>specified organism | J16.8 | Pneumonia due to other specified infectious organisms |
| 484.1 | Pneumonia in cytomegalic inclusion disease | B25.0 | Cytomegaloviral pneumonitis |
| 484.3 | Pneumonia in whooping<br>cough | A37.91<br>A37.01<br>A37.11<br>A37.81 | Whooping cough, unspecified species with pneumonia Whooping cough due to Bordetella pertussis with pneumonia Whooping cough due to Bordetella parapertussis with pneumonia Whooping cough due to other Bordetella species with pneumonia |
| 484.5 | Pneumonia in anthrax | A22.1 | Pulmonary anthrax |
| 484.6 | Pneumonia in aspergillosis | B44.0 | Invasive pulmonary aspergillosis |

| | 484.7 | Pneumonia in other systemic<br>mycoses | J17 | Pneumonia in diseases classified elsewhere |
|---|---|---|---|---|
| | 484.8 | Pneumonia in other infectious<br>diseases classified elsewhere | J17<br>B77.81 | Pneumonia in diseases classified elsewhere<br>Ascariasis pneumonia |
| | 485 | Bronchopneumonia, organism<br>unspecified | J18.0 | Bronchopneumonia, unspecified organism |
| | 486 | Pneumonia, organism<br>unspecified | J18.8<br>J18.9 | Other pneumonia, unspecified organism Pneumonia, unspecified organism |
| | 487 | Influenza with pneumonia | J10.00<br>J10.08<br>J11.00<br>J11.08<br>J12.9 | Influenza due to other identified influenza virus with unspecified type of pneumonia Influenza due to other identified influenza virus with other specified pneumonia Influenza due to unidentified influenza virus with unspecified type of pneumonia Influenza due to unidentified influenza virus with specified pneumonia Viral pneumonia, unspecified |
| | 510.x | | | Empyema |
| | 510 | Empyema with fistula | J86.0 | Pyothorax with fistula |
| | 510.9 | Empyema without mention of<br>fistula | J86.9 | Pyothorax without fistula |
| | | | J85.1 | Abscess of lung with pneumonia |
| | 136.3 | Pneumocystosis | B59 | Pneumocystosis |
| | 481 | Pneumococcal pneumonia | J13 | Pneumonia due to Streptococcus pneumoniae |
| Pneumococca<br>l | 482.9 + 041.2 | Bacterial pneumonia,<br>unspecified + pneumococcus | J15.9 + B95.3 | Unspecified bacterial pneumonia + Streptococcus pneumoniae |
| | 485 + 041.2 | Bronchopneumonia, organism<br>unspecified + pneumococcus | J18.0 + B95.3 | Bronchopneumonia, unspecified organism + Streptococcus pneumoniae |

| 486 + 041.2 | Pneumonia, organism<br>unspecified + pneumococcus | J18.8 + B95.3<br>J18.9 + B95.3 | Other pneumonia, unspecified organism + Streptococcus pneumoniae<br>Pneumonia, unspecified organism + Streptococcus pneumoniae |
|---|---|---|---|
| 510.x + 041.2 | | Em | pyema + pneumococcus |
| 510 + 041.2 | Empyema with fistula +<br>pneumococcus | J86.0 + B95.3 | Pyothorax with fistula + Streptococcus pneumoniae |
| 510.9 + 041.2 | Empyema without mention of fistula + pneumococcus | J86.9 + B95.3 | Pyothorax without fistula + Streptococcus pneumoniae |

Table 7.5 Diagnosis Codes for Identifying Pneumococcal Pneumonia and Pneumonia with Unspecified Causes

| | | ICD-9-CM | | ICD-10-CM |
|---|---|---|---|---|
| Condition | Codes | Description | Codes | Description |
| | 481 | Pneumococcal pneumonia | J13 | Pneumonia due to Streptococcus pneumoniae |
| | 482.9 +<br>041.2 | Bacterial pneumonia,<br>unspecified + pneumococcus | J15.9 + B95.3 | Unspecified bacterial pneumonia + Streptococcus pneumoniae |
| Pneumococcal | 485 + 041.2 | Bronchopneumonia, organism<br>unspecified + pneumococcus | J18.0 + B95.3 | Bronchopneumonia, unspecified organism + Streptococcus pneumoniae |
| pneumonia | 486 + 041.2 | Pneumonia, organism<br>unspecified + pneumococcus | J18.8 + B95.3<br>J18.9 + B95.3 | Other pneumonia, unspecified organism + Streptococcus pneumoniae<br>Pneumonia, unspecified organism + Streptococcus pneumoniae |
| | 510.x +<br>041.2 | | Empyema + pneumococcus | |
| | 510 + 041.2 | Empyema with fistula +<br>pneumococcus | J86.0 + B95.3 | Pyothorax with fistula + Streptococcus pneumoniae |

| | 510.9 +<br>041.2 | Empyema without mention of fistula + pneumococcus | J86.9 + B95.3 | Pyothorax without fistula + Streptococcus pneumoniae |
|---|---|---|---|---|
| | 480-486<br>487.0 | Viral, bacterial, unspecified pneumonia | | |
| | 480.9 | Viral pneumonia, unspecified | J12.9 | Viral pneumonia, unspecified |
| Pneumonia<br>with<br>unspecified | 482.9 | Bacterial pneumonia,<br>unspecified | J15.9 | Unspecified bacterial pneumonia |
| causes | 485 | Bronchopneumonia, organism<br>unspecified | J18.0 | Bronchopneumonia, unspecified organism |
| | 486 | Pneumonia, organism<br>unspecified | J18.8 | Other pneumonia, unspecified organism<br>Pneumonia, unspecified organism |
| | | | J18.9 | |

Table 7.6 Diagnosis Codes for Identifying All-Cause Pneumonia not due to HIV

| | | ICD-9-CM | | ICD-10-CM |
|---|---|---|---|---|
| Condition | Codes | Description | Codes | Description |
| | 480-486<br>487.0 | Viral, bacterial, unspecified pneumonia | | |
| All-Cause | 480 | Pneumonia due to adenovirus | J12.0 | Adenoviral pneumonia |
| An-Cause | 480.1 | Pneumonia due to respiratory<br>syncytial virus | J12.1 | Respiratory syncytial virus pneumonia |
| | 480.2 | Pneumonia due to<br>parainfluenza virus | J12.2 | Parainfluenza virus pneumonia |

| | Pneumonia due to SARS- | J12.81 | Pneumonia due to SARS-associated coronavirus |
|---|---|---|---|
| 480.3 | associated coronavirus | J12.82 | Pneumonia due to coronavirus disease 2019 |
| 480.8 | Pneumonia due to other virus<br>not elsewhere classified | J12.3<br>J12.89 | Human metapneumovirus pneumonia<br>Other viral pneumonia |
| 480.9 | Viral pneumonia, unspecified | J12.9 | Viral pneumonia, unspecified |
| 481 | Pneumococcal pneumonia<br>[Streptococcus pneumoniae<br>pneumonia] | J18.1<br>J13 | Lobar pneumonia, unspecified organism Pneumonia due to Streptococcus pneumoniae |
| 482 | Pneumonia due to Klebsiella<br>pneumoniae | J15.0 | Pneumonia due to Klebsiella pneumoniae |
| 482.1 | Pneumonia due to<br>Pseudomonas | J15.1 | Pneumonia due to Pseudomonas |
| 482.2 | Pneumonia due to Hemophilus<br>influenzae [H. influenzae] | J14 | Pneumonia due to Hemophilus influenzae |
| 482.3 | Pneumonia due to<br>Streptococcus, unspecified | J15.4 | Pneumonia due to other streptococci |
| 482.31 | Pneumonia due to<br>Streptococcus, group A | J15.4 | Pneumonia due to other streptococci |
| 482.32 | Pneumonia due to<br>Streptococcus, group B | J15.3 | Pneumonia due to streptococcus, group B |
| 482.39 | Pneumonia due to other<br>Streptococcus | J15.4 | Pneumonia due to other streptococci |
| 482.4 | Pneumonia due to<br>Staphylococcus, unspecified | J15.20 | Pneumonia due to staphylococcus, unspecified |

| 482.41 | Methicillin susceptible<br>pneumonia due to<br>Staphylococcus aureus | J15.211 | Pneumonia due to Methicillin susceptible Staphylococcus aureus |
|---|---|---|---|
| 482.42 | Methicillin resistant<br>pneumonia due to<br>Staphylococcus aureus | J15.212 | Pneumonia due to Methicillin resistant Staphylococcus aureus |
| 482.49 | Other Staphylococcus<br>pneumonia | J15.29 | Pneumonia due to other staphylococcus |
| 482.81 | Pneumonia due to anaerobes | J15.8 | Pneumonia due to other specified bacteria |
| 482.82 | Pneumonia due to escherichia<br>coli [E. coli] | J15.5 | Pneumonia due to Escherichia coli |
| 482.83 | Pneumonia due to other gram-<br>negative bacteria | J15.6 | Pneumonia due to other aerobic Gram-negative bacteria |
| 482.84 | Pneumonia due to<br>Legionnaires' disease | A48.1 | Legionnaires' disease |
| 482.89 | Pneumonia due to other<br>specified bacteria | J15.8 | Pneumonia due to other specified bacteria |
| 482.9 | Bacterial pneumonia,<br>unspecified | J15.9 | Unspecified bacterial pneumonia |
| 483.1 | Pneumonia due to chlamydia | J16.0 | Chlamydial pneumonia |
| 483.8 | Pneumonia due to other<br>specified organism | J16.8 | Pneumonia due to other specified infectious organisms |
| 484.3 | Pneumonia in whooping<br>cough | A37.91<br>A37.01<br>A37.11<br>A37.81 | Whooping cough, unspecified species with pneumonia Whooping cough due to Bordetella pertussis with pneumonia Whooping cough due to Bordetella parapertussis with pneumonia Whooping cough due to other Bordetella species with pneumonia |

| 484.5 | Pneumonia in anthrax | A22.1 | Pulmonary anthrax |
|---|---|---|---|
| | | J17 | Pneumonia in diseases classified elsewhere |
| 484.8 | Pneumonia in other infectious<br>diseases classified elsewhere | J17<br>B77.81 | Pneumonia in diseases classified elsewhere<br>Ascariasis pneumonia |
| 485 | Bronchopneumonia, organism<br>unspecified | J18.0 | Bronchopneumonia, unspecified organism |
| 486 | Pneumonia, organism<br>unspecified | J18.8<br>J18.9 | Other pneumonia, unspecified organism<br>Pneumonia, unspecified organism |
| 487 | Influenza with pneumonia | J10.00<br>J10.08<br>J11.00<br>J11.08<br>J12.9 | Influenza due to other identified influenza virus with unspecified type of pneumonia Influenza due to other identified influenza virus with other specified pneumonia Influenza due to unidentified influenza virus with unspecified type of pneumonia Influenza due to unidentified influenza virus with specified pneumonia Viral pneumonia, unspecified |
| 510.x | | | Етруета |
| 510 | Empyema with fistula | J86.0 | Pyothorax with fistula |
| 510.9 | Empyema without mention of | J86.9 | Pyothorax without fistula |
| | IIsuia | J85.1 | Abscess of lung with pneumonia |

## Table 7.7 National Drug Codes and Procedure Codes for Identifying Immunosuppressive Medications (see Excel)

Table 7.8 National Drug Codes and Procedure Codes for Identifying Influenza Vaccinations (see Excel)

Table 7.9 National Drug Codes and CPT® Codes for Identifying PPSV23 Vaccination

| Code | Type | Description |
|-------------|------|--------------|
| 90732 | CPT | Pneumovax 23 |
| 00006473900 | NDC | Pneumovax 23 |
| 00006473901 | NDC | Pneumovax 23 |
| 00006473950 | NDC | Pneumovax 23 |
| 00006474100 | NDC | Pneumovax 23 |
| 00006483701 | NDC | Pneumovax 23 |
| 00006483702 | NDC | Pneumovax 23 |
| 00006483703 | NDC | Pneumovax 23 |
| 00006489400 | NDC | Pneumovax 23 |
| 00006489400 | NDC | Pneumovax 23 |
| 00006494300 | NDC | Pneumovax 23 |
| 00006494301 | NDC | Pneumovax 23 |
| 00247040201 | NDC | Pneumovax 23 |
| 50090145200 | NDC | Pneumovax 23 |
| 50090145209 | NDC | Pneumovax 23 |
| 54569141200 | NDC | Pneumovax 23 |
| 54569653800 | NDC | Pneumovax 23 |
| 54868333901 | NDC | Pneumovax 23 |
| 54868333909 | NDC | Pneumovax 23 |
| 54868432000 | NDC | Pneumovax 23 |
| 54868432009 | NDC | Pneumovax 23 |
| 55045354202 | NDC | Pneumovax 23 |
| 00005230931 | NDC | Pnu-Imune 23 |
| 00005230933 | NDC | Pnu-Imune 23 |
| 54868070700 | NDC | Pnu-Imune 23 |

Table 7.10 National Drug Codes and CPT® Codes for Identifying Recombinant Zoster Vaccination

| Code | Type | Description |
|-------------|------|-------------|
| 58160082801 | NDC | Shingrix |
| 58160082803 | NDC | Shingrix |
| 50090514700 | NDC | Shingrix |
| 58160081912 | NDC | Shingrix |
| 58160082311 | NDC | Shingrix |

| 50090337200 | NDC | Shingrix |
|-------------|-----|--------------------------|
| 90750 | CPT | Zoster Vaccine |
| | | Recombinant, Adjuvanted, |
| | | Suspension for |
| | | Intramuscular Injection |

## Table 7.11 CPT® Codes to Identify CD4 Laboratory Tests

| Code | Туре | Description |
|-------|------|----------------------|
| 86361 | CPT | Absolute CD4 count |
| 86360 | CPT | Absolute CD4 and CD8 |
| | | counts with ratio |

## Table 7.12 CPT® Codes to identify Viral Load Laboratory Tests

| Code | Type | Description |
|---|---|---|
| 87534 | CPT | Infectious agent detection by<br>nucleic acid (DNA or RNA);<br>HIV-1, direct probe technique |
| 87535 | CPT | Infectious agent detection by<br>nucleic acid (DNA or RNA);<br>HIV-1, amplified probe<br>technique |
| 87536 | CPT | Infectious agent detection by<br>nucleic acid (DNA or RNA);<br>HIV-1, quantification |

Table 7.13 National Drug Codes for Identifying Candidiasis Antifungals (see Excel)

## **Document Approval Record**

| Document Name: | B1851217 FINAL STATISTICAL ANALYSIS PLAN V1.3_07Dec2023 |
|-----------------|---------------------------------------------------------|
| Document Title: | B1851217 FINAL STATISTICAL ANALYSIS PLAN V1.3_07Dec2023 |

| Signed By: | Date(GMT) | Signing Capacity |
|------------|----------------------|---------------------|
| PPD | 11-Dec-2023 18:07:25 | Contributing Author |
| | 11-Dec-2023 18:55:58 | Manager Approval |